CLINICAL TRIAL: NCT00001864
Title: Amblyopia Treatment Study
Brief Title: Amblyopia (Lazy Eye) Treatment Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990110; 99-EI-0110
Record Dates: First submitted 1999-11-03; First posted 2002-05-22 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-11

CONDITIONS: Amblyopia; Anisometropia; Strabismus
Keywords: Lazy Eye; Atropine Penalization; Patching; Vision Loss; Amblyopia
MeSH Terms: conditions — Amblyopia; Anisometropia; Strabismus; Vision Disorders | interventions — Atropine; Transdermal Patch

INTERVENTIONS:
Drug: Atropine
Device: Patch

SUMMARY:
The purpose of this study is to compare the results of two standard treatments for amblyopia in order to find out if one is more effective than the other. Amblyopia, which develops in childhood, is also called "lazy eye," because one eye is not being used properly. The brain favors the other eye for some reason, such as crossing or turning out of the eyes, and vision in the weak eye is reduced.

Amblyopia is treated by forcing the child to use the weak eye. There are two ways to do this: 1) a patch placed over the "good" eye forces the child to use the weak eye; or 2) an eye drop placed in the "good" eye once a day to blur vision in that eye makes the child rely on the weak eye. The success rates with both of these methods have been reported to be about the same; this study will try to identify if one is more effective than the other.

Children will be randomly assigned by computer to one of the following two treatment methods:

Patch

The child initially will wear a patch over the "good" eye for 8 to 12 hours every day. If vision in the weak eye improves, the patching time will be decreased. If vision remains good after 3 months, the patching will be stopped, unless the child's doctor believes treatment should continue. If vision in the weak eye does not improve, the patching time will be increased.

Eye Drops

The child will be given one drop per day of atropine in the "good" eye. If vision in the weak eye improves, the drops will be given less often. If the vision remains good after 3 months, the drops will be stopped, unless the child's doctor believes treatment should continue. If the initial daily drop does not improve the vision in the weak eye, the child's eyeglasses may be changed to try to further blur the vision in the "good" eye.

After 6 months, treatment may be stopped if it has not been successful. If treatment has been successful after 6 months, it may be continued at a reduced amount or stopped.

Follow-up visits will be scheduled every 4 weeks for the first 6 months and every 2 to 4 months after that until the end of the 2-year study. During each visit the eyes will be examined for eye movements and vision, and the pupils will be dilated to examine the inside of the eye.

DETAILED DESCRIPTION:
The Amblyopia Treatment Study (ATS) has been designed as a randomized, controlled single-masked multi-center clinical trial with the following objectives:

To determine whether the success rate with atropine treatment of amblyopia due to strabismus or anisometropia in patients less than 7 years old is equivalent to the success rate with occlusion (patching) therapy.

To develop more precise estimates of the success rates of amblyopia treatment.

To identify factors that may be associated with successful treatment of amblyopia.

To collect data on the clinical course of treated amblyopia to provide more precise estimates of treatment kinetics than now available.

ELIGIBILITY:
Age less than 7 years.

Able to measure surrounded single optotype visual acuity using the ATS BVAT protocol.

Amblyopia associated with strabismus (comitant or incomitant), anisometropia, or both.

No more than 2 months of amblyopia therapy in the past 2 years.

No current vision therapy or orthoptics.

Visual acuity in the sound eye greater than or equal to 20/40.

Visual acuity in the amblyopic eye less than or equal to 20/40 and greater than or equal to 20/100.

Inter-eye acuity difference (IAD) greater than or equal to 3 LogMAR lines.

No ocular cause for reduced visual acuity.

Cycloplegic refraction and ocular examination within 2 months of enrollment.

No myopia.

Hyperopic/astigmatic refractive error, if present, corrected for at least 4 weeks.

No prior intraocular surgery.

Downs Syndrome not present.

No known skin reactions to patch or bandage adhesives.

No known allergy to atropine or other cycloplegics.

Availability for at least 6 months of follow-up, has a home phone (or access to phone), and willing to be contacted by Jaeb Center staff.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1999-05; Study Completion 2001-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Woodruff G, Hiscox F, Thompson JR, Smith LK. Factors affecting the outcome of children treated for amblyopia. Eye (Lond). 1994;8 ( Pt 6):627-31. doi: 10.1038/eye.1994.157. PMID 7867817
- [Background] Shaw DE, Fielder AR, Minshull C, Rosenthal AR. Amblyopia--factors influencing age of presentation. Lancet. 1988 Jul 23;2(8604):207-9. doi: 10.1016/s0140-6736(88)92301-x. PMID 2899674
- [Background] Simons K. Preschool vision screening: rationale, methodology and outcome. Surv Ophthalmol. 1996 Jul-Aug;41(1):3-30. doi: 10.1016/s0039-6257(97)81990-x. PMID 8827927